CLINICAL TRIAL: NCT04177212
Title: Prospective, Multicenter, Parallel-group, Evaluator-blind, Randomized Study to Investigate the Effectiveness and Safety of MRZF111 in the Treatment of décolleté Wrinkles
Brief Title: Investigation of the Effectiveness and Safety of MRZF111 in the Treatment of Décolleté Wrinkles
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Merz Aesthetics GmbH (Industry)
Collaborators: Merz Pharmaceuticals GmbH (Industry)
Responsible Party: Sponsor
Organization: Merz North America, Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: M930521001
Record Dates: First submitted 2019-11-20; First posted 2019-11-26 (Actual); Results first posted 2023-12-26 (Actual); Last update posted 2023-12-26 (Actual); Status verified 2023-12

CONDITIONS: Décolleté Wrinkles

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (2):
- 3 MRZF111 injection cycles (Experimental): Enrolled subjects will receive 3 injection cycles in total at time points Day 1, Week 8, and Week 16.
  Interventions: Device: MRZF111
- 2 MRZF111 injection cycles (Experimental): Enrolled subjects will receive 2 injection cycles in total at time points Day 1, and Week 16.
  Interventions: Device: MRZF111

INTERVENTIONS:
Device: MRZF111 — MRZF111 kit consisting of one syringe of RADIESSE® Volume injectable implant, injection needles and additional components. Physiological saline solution (0.9% NaCl) is used to dilute Radiesse Volume by 1:2. Radiesse consists of calcium hydroxylapatite particles suspended in an aqueous-based gel carrier.
  Other Names: Radiesse

SUMMARY:
To evaluate the effectiveness and safety of MRZF111 treatment for improvement of décolleté wrinkles as assessed on the Merz Aesthetics Scales (MAS) Décolleté Wrinkles-At Rest.

ELIGIBILITY:
Inclusion Criteria:

* Female between ≥18 and ≤65 years old.
* Décolleté wrinkles with a rating of moderate to severe (grade 2 to 3) on the MAS Décolleté Wrinkles-At Rest as determined by the blinded live rater and confirmed by the treating investigator afterwards.

Exclusion Criteria:

* Any previous treatment with fat injections, poly L-lactic acid or permanent dermal fillers (e.g., silicone, polymethyl methacrylate) in the décolleté.
* Any previous surgery, including plastic surgery, or surgical permanent implant in the décolleté or in the breasts that could interfere with effectiveness and safety.
* Any previous thread lifting in the décolleté.
* Previous treatment with collagen fillers, calcium hydroxylapatite (CaHa), and/or long-lasting hyaluronic acid (HA) fillers (e.g., Belotero® Intense/Volume, Juvéderm® Volift/Volbella) in the décolleté within the past 24 months before baseline.
* Previous treatment with other HA fillers in the décolleté within the past 12 months before baseline.
* Previous treatment with botulinum toxin, ablative or fractional laser, microdermabrasion, microneedling, chemical peels and/or non-invasive skin tightening (e.g., ultrasound, radiofrequency, intense pulsed light treatment) in the décolleté within the past 6 months before baseline.

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 117 (Actual)
Dates: Start 2019-12-04 (Actual); Primary Completion 2020-11-17 (Actual); Study Completion 2021-02-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Merz Medical Expert, Study Director — Merz North America, Inc.
Locations (9):
- Germany (9):
  - Merz Investigational Site #0490189, Bad Soden
  - Merz Investigational Site #0490375, Drensteinfurt
  - Merz Investigational Site #0490095, Hamburg
  - Merz Investigational Site #0490345, Hamburg
  - Merz Investigational Site #0490309, Kassel
  - Merz Investigational Site #0490371, München
  - Merz Investigational Site #0490372, München
  - Merz Investigational Site #0490362, Potsdam
  - Merz Investigational Site #0490367, Wuppertal

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at 9 investigational sites in Germany from 04 December 2019 to 23 February 2021. A total of 117 participants were enrolled and randomized in the study, out of which 90 participants completed the study.
Pre-assignment Details: Primary effectiveness analysis was done on pooled data.Further supportive explorative analyses done separately by Groups A and B for primary effectiveness outcome measure(OM) and for secondary effectiveness OM 2,but this analysis was not part of main primary effectiveness analysis.As per planned analysis based on protocol and SAP,data for secondary effectiveness outcome measures(3 to 6)were planned to be analyzed for pooled treatment groups,hence pooled data reported for these outcome measures.
Groups:
- Group A: MRZF111 (3 Injections): Participants received three injections of MRZF111, a subdermal injection in the central part of the décolleté area on Day 1, Week 8, and Week 16. Participants received a total volume of 13.5 milliliter (mL) MRZF111 over the complete course of treatment.
- Group B: MRZF111 (2 Injections): Participants received two injections of MRZF111, a subdermal injection in the central part of the décolleté area on Day 1 and Week 16. Participants received a total volume of 9.0 mL MRZF111 over the complete course of treatment.
Period: Overall Study
Arm/Group | Group A: MRZF111 (3 Injections) | Group B: MRZF111 (2 Injections)
Started | 55 | 62
Safety Analysis Set (Participants who were randomized to Group A but treated according to the injection scheme of Group B due to coronavirus disease 2019 (COVID-19) pandemic measures were analyzed in Group B. Participants who were treated only once due to any reason were analyzed in Group B.) | 43 | 74
Modified Full Analysis Set (Participants randomized to Group A but treated as per Group B injection scheme due to COVID-19 pandemic measures were analyzed in Group B. Participants treated only once with all missing treatments due to reasons not related to pandemic measures such as premature withdrawal/protocol deviations, were analyzed in treatment group they were randomized to and participants treated only once with at least one missing treatment due to reasons related to pandemic measures were analyzed in Group B.) | 46 | 71
Completed | 43 | 47
Not Completed | 12 | 15
Not completed — Withdrawal by Subject | 9 | 7
Not completed — Due to COVID-19 Pandemic | 1 | 2
Not completed — Physician Decision | 1 | 0
Not completed — Lost to Follow-up | 0 | 3
Not completed — Adverse Event | 0 | 1
Not completed — Other | 1 | 2

BASELINE CHARACTERISTICS:
Population: The safety analysis set (SAS) included participants who were randomized to Group A but treated according to the injection scheme of Group B due to COVID-19 pandemic measures and were analyzed in Group B. Participants who were treated only once were analyzed in Group B.
Groups:
- Group A: MRZF111 (3 Injections): Participants received three injections of MRZF111, a subdermal injection in the central part of the décolleté area on Day 1, Week 8, and Week 16. Participants received a total volume of 13.5 mL MRZF111 over the complete course of treatment.
- Total: Total of all reporting groups
Arm/Group | Group A: MRZF111 (3 Injections) | Group B: MRZF111 (2 Injections) | Total
Number analyzed (Participants) | 43 | 74 | 117
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.2 (6.0) | 52.8 (7.3) | 53.0 (6.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 43 | 74 | 117
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 43 | 74 | 117
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kilogram per square meter (kg/m^2)] | 24.0 (3.9) | 23.8 (3.4) | 23.9 (3.5)

OUTCOME MEASURES:

1. Primary Outcome: Responder Rate for Décolleté Wrinkles According to the Merz Aesthetics Scale (MAS)-At Rest Scale as Assessed by the Blinded Live Rater
Description: The percentage of responders (responder rate) was defined as greater than or equal to (>=) 1-point improvement on MAS décolleté wrinkles from baseline to 16 weeks after last treatment as assessed by the blinded live rater. Responder rate for décolleté wrinkles at rest was assessed using MAS-at rest scale. The MAS-at rest scale included five-point scale: 0 = no wrinkles, 1 = mild wrinkles, 2 = moderate wrinkles, 3 = severe wrinkles, 4 = very severe wrinkles. The higher score indicated the worst outcome.
Time Frame: 16 weeks after the last treatment on Week 16 (at Week 32)
Population: The modified full analysis set (FAS) included participants who were treated at least once. Here, overall number of participants analyzed signifies participants who were evaluable for this outcome measure. Modified FAS (observed cases) was used for Groups A and B. Modified FAS (missing data imputed via multiple imputation approach) was used for pooled treatment group.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Pooled Treatment Group (Group A: MRZF111 [3 Injections] + Group B: MRZF111 [2 Injections]): Participants received MRZF111 subdermal injection in the central part of the décolleté area (Group A: three injections on Day 1, Week 8, and Week 16; Group B: two injections on Day 1 and Week 16). Participants received a total volume of 13.5 mL (Group A) or 9.0 mL (Group B) MRZF111 over the complete course of treatment.
Arm/Group | Group A: MRZF111 (3 Injections) | Group B: MRZF111 (2 Injections) | Pooled Treatment Group (Group A: MRZF111 [3 Injections] + Group B: MRZF111 [2 Injections])
Number analyzed (Participants) | 39 | 49 | 117
percentage of participants | 71.8 [56.2 to 83.5] | 83.7 [71.0 to 91.5] | 73.5 [62.8 to 82.5]
Statistical Analysis 1: Comparison: Pooled Treatment Group (Group A: MRZF111 [3 Injections] + Group B: MRZF111 [2 Injections]); Between Groups calculation were not done because comparing Groups A and B was not part of the objective of this investigation; Test type: Other; p < 0.0001, One-sided binomial test — P-value for testing null-hypothesis that response of Pooled Group was less or equal to 50 percent (%)

2. Secondary Outcome: Responder Rate for Décolleté Wrinkles According to the MAS-Dynamic Scale as Assessed by the Blinded Live Rater (Last Observation Carried Forward [LOCF])
Description: The percentage of responders (responder rate) was defined as >= 1-point improvement on MAS décolleté wrinkles from baseline to 16 weeks after last treatment as assessed by the blinded live rater. Responder rate for décolleté wrinkles at dynamic was assessed using MAS-Dynamic Scale. The MAS-Dynamic Scale included five-point scale: 0 = no wrinkles, 1 = mild wrinkles, 2 = moderate wrinkles, 3 = severe wrinkles, 4 = very severe wrinkles. The higher score indicated the worst outcome.
Time Frame: 16 weeks after the last treatment on Week 16 (at Week 32)
Population: The modified FAS included participants who were treated at least once. Here, overall number of participants analyzed signifies participants who were evaluable for this outcome measure. Modified FAS (observed cases) was used for Groups A and B. Modified FAS (missing data imputed with LOCF) was used for pooled treatment group.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Group A: MRZF111 (3 Injections) | Group B: MRZF111 (2 Injections) | Pooled Treatment Group (Group A: MRZF111 [3 Injections] + Group B: MRZF111 [2 Injections])
Number analyzed (Participants) | 39 | 49 | 117
percentage of participants | 74.4 [58.9 to 85.4] | 69.4 [55.5 to 80.5] | 65.8 [56.8 to 73.8]
Statistical Analysis 1: Comparison: Pooled Treatment Group (Group A: MRZF111 [3 Injections] + Group B: MRZF111 [2 Injections]); [analysis description as in outcome 1, analysis 1]; Test type: Other; p = 0.0003, One-sided binomial test — P-value for testing null-hypothesis that response of Pooled Group was less or equal to 50%

3. Secondary Outcome: Percentage of Participants With Aesthetic Improvement After the Décolleté Wrinkles Treatments Based on Investigator's Treatment Satisfaction Assessment Scale (LOCF)
Description: Treatment satisfaction is defined as a rating of +3 (Very satisfied), +2 (Satisfied) or +1 (Somewhat satisfied). The treating investigators were asked to rate their level of satisfaction with the aesthetic appearance of the participant's décolleté after treatment. The investigator responded on a 7-point scale: - 3 = very dissatisfied, - 2 = dissatisfied, - 1 = somewhat dissatisfied, 0 = neither satisfied nor dissatisfied, + 1 = somewhat satisfied, + 2 = satisfied, + 3 = very satisfied. The higher score indicated aesthetic improvement.
Time Frame: 16 weeks after the last treatment on Week 16 (at Week 32)
Population: The modified pooled FAS included participants who were treated at least once. As per the planned analysis based on protocol and SAP, this secondary effectiveness outcome measure was planned to be analyzed for the pooled treatment groups as Groups A and B comparison was not objective of this investigation, hence pooled data was reported for this secondary outcome measure.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Pooled Treatment Group (Group A: MRZF111 [3 Injections] + Group B: MRZF111 [2 Injections])
Number analyzed (Participants) | 117
percentage of participants | 76.9 [68.5 to 83.6]

4. Secondary Outcome: Percentage of Participants With Aesthetic Improvement After the Décolleté Wrinkles Treatments Based on Participant's Treatment Satisfaction Assessment Scale (LOCF)
Description: Treatment satisfaction is defined as a rating of +3 (Very satisfied), +2 (Satisfied) or +1 (Somewhat satisfied). The participants were asked to rate their level of satisfaction with the aesthetic appearance of their décolleté after treatment. The participants responded on a 7-point scale: - 3 = very dissatisfied, - 2 = dissatisfied, - 1 = somewhat dissatisfied, 0 = neither satisfied nor dissatisfied, + 1 = somewhat satisfied, + 2 = satisfied, + 3 = very satisfied. The higher score indicated aesthetic improvement.
Time Frame: 16 weeks after the last treatment on Week 16 (at Week 32)
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Pooled Treatment Group (Group A: MRZF111 [3 Injections] + Group B: MRZF111 [2 Injections])
Number analyzed (Participants) | 117
percentage of participants | 70.1 [61.3 to 77.6]

5. Secondary Outcome: Percentage of Participants With Global Aesthetic Improvement Based on the Investigator's Global Aesthetic Improvement Scale on Décolleté Wrinkles (iGAIS-Wrinkles) as Assessed by the Treating Investigator (LOCF)
Description: Improvement is defined as a rating of +1 (Improved), +2 (Much improved) or +3 (Very much improved). Treating investigators used iGAIS-Wrinkles to assess aesthetic improvement in participants. The assessment was performed by treating investigator by live rating using standardized pre-treatment photographs for comparison. Treating investigator was asked based on their clinical experience to rate their overall impression of change of participant's décolleté wrinkles due to treatment. The investigator responded on a 7-point scale: - 3 = very much worse, - 2 = much worse, - 1 = worse, 0 = no change, + 1 = improved, + 2 = much improved, + 3 = very much improved. Higher score indicated aesthetic improvement.
Time Frame: 16 weeks after the last treatment on Week 16 (at Week 32)
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Pooled Treatment Group (Group A: MRZF111 [3 Injections] + Group B: MRZF111 [2 Injections])
Number analyzed (Participants) | 117
percentage of participants | 78.6 [70.4 to 85.1]

6. Secondary Outcome: Percentage of Participants With Global Aesthetic Improvement Based on the Subject's Global Aesthetic Improvement Scale on Décolleté Wrinkles (sGAIS-Wrinkles) as Assessed by the Participant (LOCF)
Description: Improvement is defined as a rating of +1 (Improved), +2 (Much improved) or +3 (Very much improved). The sGAIS-wrinkles was used to assess aesthetic improvement in the participants. The assessment was performed by the participant by live rating using standardized pre-treatment photographs for comparison. The participant was asked to rate their overall impression of change of their décolleté wrinkles due to treatment. The participant responded on a 7-point scale: - 3 = very much worse, - 2 = much worse, - 1 = worse, 0 = no change, + 1 = improved, + 2 = much improved, + 3 = very much improved.
Time Frame: 16 weeks after the last treatment on Week 16 (at Week 32)
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Pooled Treatment Group (Group A: MRZF111 [3 Injections] + Group B: MRZF111 [2 Injections])
Number analyzed (Participants) | 117
percentage of participants | 66.7 [57.7 to 74.6]

7. Secondary Outcome: Percentage of Participants With at Least One Treatment-related Treatment-emergent Adverse Event (TEAE)
Time Frame: Up to Week 52
Population: SAS included participants who were randomized to Group A but treated according to the injection scheme of Group B due to COVID-19 pandemic measures and were analyzed in Group B. Participants who were treated only once were analyzed in Group B.
Measure: Number; unit: percentage of participants
Arm/Group | Group A: MRZF111 (3 Injections) | Group B: MRZF111 (2 Injections)
Number analyzed (Participants) | 43 | 74
percentage of participants | 51.2 | 31.1

ADVERSE EVENTS:
Time Frame: Up to Week 52
Description: The investigator reported adverse events systematically at each visit.
Arm/Group | Group A: MRZF111 (3 Injections) | Group B: MRZF111 (2 Injections)
All-Cause Mortality (participants affected / at risk) | 0/43 | 0/74
Serious Adverse Events (participants affected / at risk) | 4/43 | 5/74
Other Adverse Events (participants affected / at risk) | 21/43 | 25/74
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Group A: MRZF111 (3 Injections) (N=43) | Group B: MRZF111 (2 Injections) (N=74)
Ankle fracture (Injury, poisoning and procedural complications) | 1 | 0
Concussion (Injury, poisoning and procedural complications) | 1 | 0
Contusion (Injury, poisoning and procedural complications) | 1 | 0
Meniscus injury (Injury, poisoning and procedural complications) | 0 | 1
Post-traumatic neck syndrome (Injury, poisoning and procedural complications) | 1 | 0
Stress fracture (Injury, poisoning and procedural complications) | 0 | 1
Breast cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Keratoacanthoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Superficial spreading melanoma stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Facial paralysis (Nervous system disorders) | 0 | 1
Vaginal haemorrhage (Reproductive system and breast disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Group A: MRZF111 (3 Injections) (N=43) | Group B: MRZF111 (2 Injections) (N=74)
Injection site haematoma (General disorders) | 12 | 7
Injection site pain (General disorders) | 4 | 13
Injection site erythema (General disorders) | 3 | 8
Injection site discolouration (General disorders) | 6 | 3
Injection site nodule (General disorders) | 3 | 3
Nasopharyngitis (Infections and infestations) | 4 | 10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Publication of study information usually requires agreement with the sponsor. In case of justified doubts by the sponsor, the INVESTIGATOR will consider these doubts in the publication as long as the scientific neutrality is not affected.

DOCUMENTS (2):
  • Study Protocol (2023-09-05): https://cdn.clinicaltrials.gov/large-docs/12/NCT04177212/Prot_000.pdf
  • Statistical Analysis Plan (2023-09-05): https://cdn.clinicaltrials.gov/large-docs/12/NCT04177212/SAP_001.pdf